CLINICAL TRIAL: NCT03572478
Title: A Phase Ib/IIa Study of Rucaparib (PARP Inhibitor) Combined With Nivolumab in Metastatic Castrate - Resistant Prostate Cancer and Advanced/Recurrent Endometrial Cancer
Brief Title: Rucaparib and Nivolumab in Patients With Prostate or Endometrial Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to lack of efficacy.
Sponsor: University of Chicago (Other)
Collaborators: Bristol-Myers Squibb (Industry); Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-0154
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Results first posted 2021-02-12 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer; Endometrial Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Endometrial Neoplasms | interventions — rucaparib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Combination Therapy (Phase 1b Cohort) (Experimental): Participants will receive rucaparib plus nivolumab in 4 week cycles.
  Interventions: Drug: Rucaparib; Drug: Nivolumab
- Rucaparib (Phase 2b Randomized Cohort) (Experimental): Participants randomized to receive rucaparib alone in 4 week cycles.
  Interventions: Drug: Rucaparib
- Nivolumab (Phase 2b Randomized Cohort) (Experimental): Participants randomized to receive nivolumab alone in 4 week cycles.
  Interventions: Drug: Nivolumab
- Combination Therapy (Phase 2b Randomized Cohort) (Experimental): Participants randomized to receive rucaparib plus nivolumab in 4 week cycles. Participants will receive rucaparib alone in cycle 1 and begin nivolumab on day 1 of Cycle 2.
  Interventions: Drug: Rucaparib; Drug: Nivolumab

INTERVENTIONS:
Drug: Rucaparib — 600 mg taken by mouth twice daily.
  Other Names: Rubraca(R)
  Arms: Combination Therapy (Phase 1b Cohort); Combination Therapy (Phase 2b Randomized Cohort); Rucaparib (Phase 2b Randomized Cohort)
Drug: Nivolumab — 480 mg given by intravenous (IV) infusion every 4 weeks.
  Other Names: Opdivo(R)
  Arms: Combination Therapy (Phase 1b Cohort); Combination Therapy (Phase 2b Randomized Cohort); Nivolumab (Phase 2b Randomized Cohort)

SUMMARY:
This is a phase 1/phase 2a study of the combination of immune checkpoint inhibitor (nivolumab) in combination with the PARP inhibitor (rucaparib) for patients with metastatic castration resistant prostate cancer (mCRPC) and metastatic/recurrent endometrial cancer.

In the phase 1 portion, the safety of the combination dosing will be determined. If the combination dosing is determined to be safe and feasible, the study will move onto phase 2a.

In the phase 2a portion, participants will be randomized to receive either: rucaparib alone, nivolumab alone, or combination therapy (rucaparib and nivolumab).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and the willingness to signed a written informed consent document.
* Patients must have histologically or cytologically confirmed CRPC or endometrial cancer that is metastatic. Evidence of disease progression on a prior therapy is not required.
* Patients must have at least one lesion that is amenable to biopsy and the treating physician must deem this safe.
* Patient must be willing to undergo two mandatory research-only biopsies.
* Prostate cancer patients:

  * Patients must be surgically or medically castrated, with serum testosterone levels ≤ 50 ng/mL Patients being treated with Gonadotropin-releasing hormone (GnRH) agonists must have such therapy continued throughout the study.
  * Patients should have received at least one androgen receptor (AR)-targeted therapy with abiraterone acetate or enzalutamide. Multiple lines of prior AR-targeted therapy and chemotherapy are permitted. A washout of two weeks from prior endocrine therapy (other than GnRH agonist); four weeks washout period from prior cytotoxic chemotherapy or other anticancer agents is required (prior to day 1 of study therapy); six weeks washout period to allow for anti-androgen withdrawal for patients managed with antiandrogen therapy such as bicalutamide.
* Endometrial cancer patients:

  * An unlimited number of prior hormonal and/or chemotherapy regimens are permitted. A washout of two weeks from prior endocrine therapy (other than GnRH agonist) and four weeks from prior cytotoxic chemotherapy or other anticancer agents is required (prior to day 1 of study therapy).
* At least 5 days should have elapsed since any non-study related minor surgical procedure and at least 21 days since any major surgical procedure prior to the first dose of rucaparib and the first dose of nivolumab.
* Must have an ability to swallow pills or capsules. Patients should have no current clinical evidence of bowel obstruction.
* Age must be ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status must be ≤ 1
* Patients must have normal hepatic, renal and marrow function as defined below:

  * hemoglobin > 10 g/dL
  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 150,000/mcL
  * total bilirubin within normal institutional limits
  * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Prior palliative radiotherapy must have been completed at least 2 weeks prior to first dose of study drug. Subjects with symptomatic tumor lesions at baseline that may require palliative radiotherapy within 4 weeks of first dose of study drug are strongly encouraged to receive palliative radiotherapy prior to enrollment.
* Reproductive Status: Rucaparib caused post-implantation loss (100% early resorptions) at all doses administered in an embryo-fetal development study. Based on its mechanism of action, nivolumab can cause fetal harm when administered to a pregnant woman. Pregnant women are therefore not eligible for this study.

  * Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test result less than 3 days prior to administration of the first dose of rucaparib.
  * WOCBP must not be considering getting pregnant during the study.
  * WOCBP and their male partners must agree to use a highly effective, reliable form of contraception during treatment; for 6 months following the last dose of rucaparib; and for at least 5 months following the last dose of nivolumab.
  * Men who are sexually active with WOCBP must agree to use a highly effective, reliable form of contraception during treatment; 6 months following the last dose of rucaparib; and for a period of 7 months after the last dose of nivolumab .
  * In addition to the above methods of contraception, use of a condom by male patients is recommended to prevent transfer of drug through semen.

Exclusion Criteria:

* Patients with active, known, or suspected autoimmune disease. Subjects with vitiligo, type I diabetes, mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, childhood asthma that is not currently active, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration except for adrenal replacement steroid doses > 10 mg daily prednisone equivalent in the absence of active autoimmune disease. Note: Treatment with a short course of steroids (< 5 days) up to 7 days prior to initiating study drug is permitted.
* Patients who are receiving any other investigational agents.
* Prior exposure to PD-1 or PD-L1 inhibitors, other immune checkpoint inhibitors (e.g. anti-LAG-3, and anti-CTLA-4 antibodies), or PARP inhibitors.
* Patients with a "currently active" second invasive malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and have been free of disease for ≥ 1 years.
* Patients with known and untreated or progressing brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients whose brain metastases have been treated with surgery and/or radiotherapy and are without evidence of progression on scan for at least 4 weeks, and are off steroids or antiseizure medications, will be eligible .
* Patients with symptomatic or impending spinal cord compression are not eligible unless appropriately treated.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab or rucaparib.
* Based on in vitro CYP interaction studies, caution should be used for concomitant medications with a narrow therapeutic window that are substrates of CYP2C19, CYP2C9, and/or CYP3A. Selection of an alternate concomitant medication is recommended. Caution should also be exercised for concomitant use of certain statin drugs (e.g. rosuvastatin and fluvastatin) due to potential increase in exposure from inhibition of BCRP and CYP2C9. An updated list of clinically relevant P450 drug interactions (e.g: Flockhart Table http://medicine.iupui.edu/clinpharm/ddis/main-table/) should be reviewed while screening patients for study.

  * Patients taking warfarin should have international normalized ration (INR) monitored regularly according to standard institutional practices
  * Because rucaparib is a moderate inhibitor of P-gp in vitro, caution should be exercised for patients receiving rucaparib and requiring concomitant medication with digoxin. Patients taking digoxin should have their digoxin levels monitored after starting rucaparib and then regularly per standard clinical practice.
* Patients on parenteral nutrition are not eligible. Patients must not have a pre-existing duodenal stent or any gastrointestinal disorder or defect that would, in the opinion of the treating investigator, interfere with absorption of rucaparib.
* Uncontrolled intercurrent illness including, but not limited to, requirement for oxygen therapy, ongoing or active infection other than minor urinary tract infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known history of chronic hepatitis B or C as evidenced by:

  * Positive test for hepatitis B surface antigen
  * Positive test for qualitative hepatitis C viral load (by polymerase chain reaction [PCR])
  * Note: Subjects with positive hepatitis C antibody and negative quantitative hepatitis C by polymerase chain reaction (PCR) are eligible.
* Human Immunodeficiency Virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with rucaparib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Prior organ allograft or allogeneic bone marrow transplantation.
* Adverse effect of prior therapy not improved to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or below with the exception of alopecia or lymphopenia. Ongoing Grade 2 non-hematologic toxicity (e.g. neuropathy) related to most recent treatment regimen may be permitted with prior advanced approval from the Lead Principal Investigator.
* Initiated denosumab or bisphosphonate therapy or adjusted denosumab or bisphosphonate dose/regimen within 4 weeks prior to first dose of rucaparib. Patients on a stable denosumab or bisphosphonate regimen are eligible and may continue treatment.
* Evidence or history of active or latent tuberculosis infection including purified protein derivative (PPD) recently converted to positive.
* Use of non-oncology vaccines containing live virus for prevention of infectious diseases within 12 weeks prior to study drug. The use of inactivated seasonal influenza vaccines, e.g., Fluzone®, will be permitted on study without restriction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated due to lack of efficacy such that participants were enrolled only in phase 1 cohort (single arm).
Groups:
- Combination Therapy (Phase 1 Cohort): Although we initially planned to conduct phase 1/2a study in the protocol, participants were enrolled only in phase 1 cohort.
  Participants will receive rucaparib plus nivolumab in 4 week cycles.
  Rucaparib: 600 mg taken by mouth twice daily.
  Nivolumab: 480 mg given by intravenous (IV) infusion every 4 weeks.
Period: Overall Study
Arm/Group | Combination Therapy (Phase 1 Cohort)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy (Phase 1 Cohort)
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 72 [60 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose Limiting Toxicities (DLT) (Phase 1)
Description: Dose limiting toxicities (DLT) is measured by patients with grade 3 or 4 toxicity within 4 weeks of starting leading to discontinuation of rucaparib for at least 1 week
Time Frame: 8 weeks
Population: Two patients were not evaluable for DLT due to rapidly progressive disease.
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy (Phase 1 Cohort)
Number analyzed (Participants) | 10
percentage of participants | 50

2. Primary Outcome: Frequency of Patients With T Cell Inflammation in the Tumor Compared Between Treatment Arms (Phase 2)
Time Frame: 4 weeks
Population: No participants were enrolled in Phase 2 cohort.
Arm/Group | Combination Therapy (Phase 1 Cohort)
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Disease Progression in Prostate Cancer Patients (Phase 2)
Time Frame: 24 months
Population: No participants were enrolled in Phase 2 cohort.
Arm/Group | Combination Therapy (Phase 1 Cohort)
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Disease Progression in Endometrial Cancer Patients (Phase 2)
Time Frame: 24 months
Population: No participants were enrolled in Phase 2 cohort.
Arm/Group | Combination Therapy (Phase 1 Cohort)
Number analyzed (Participants) | 0

5. Secondary Outcome: Response Rate in Prostate Cancer Patients (Phase 2)
Time Frame: 24 months
Population: No participants were enrolled in Phase 2 cohort.
Arm/Group | Combination Therapy (Phase 1 Cohort)
Number analyzed (Participants) | 0

6. Secondary Outcome: Response Rate in Endometrial Cancer Patients (Phase 2)
Time Frame: 24 months
Population: No participants were enrolled in Phase 2 cohort.
Arm/Group | Combination Therapy (Phase 1 Cohort)
Number analyzed (Participants) | 0

7. Secondary Outcome: Changes in Number of T Cells in Tumor Samples Compared Between Treatment Arms (Phase 2)
Time Frame: 4 weeks
Population: No participants were enrolled in Phase 2 cohort.
Arm/Group | Combination Therapy (Phase 1 Cohort)
Number analyzed (Participants) | 0

8. Secondary Outcome: Correlation of Change in T Cells in Tumor Samples and PTEN Mutation Status (Phase 2)
Time Frame: 4 weeks
Population: No participants were enrolled in Phase 2 cohort.
Arm/Group | Combination Therapy (Phase 1 Cohort)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 28 days after the end of treatment
Arm/Group | Combination Therapy (Phase 1 Cohort)
All-Cause Mortality (participants affected / at risk) | 7/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy (Phase 1 Cohort) (N=12)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
anorexia (Metabolism and nutrition disorders) | 1
neoplasms benign, malignant and unspecified (Nervous system disorders) | 1
anemia (Blood and lymphatic system disorders) | 1
acute kidney injury (Renal and urinary disorders) | 1
death (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy (Phase 1 Cohort) (N=12)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 5
Anemia (Blood and lymphatic system disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase increased (Investigations) | 8
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema limbs (General disorders) | 2
Esophageal obstruction (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 7
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lymphocyte count decreased (Investigations) | 4
Lymphocyte count increased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 7
Neutrophil count decreased (Investigations) | 2
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT03572478/Prot_SAP_000.pdf